CLINICAL TRIAL: NCT00203073
Title: A Multi-Center, Randomized, Open Label Study To Evaluate Safety, Tolerability And Efficacy Of Treatment With Mitoxantrone; Pre-Treatment With Glatiramer Acetate (GA) Versus Treatment With GA Alone In Relapsing Forms Of Multiple Sclerosis.
Brief Title: A Study to Evaluate the Safety and Effectiveness of Novantrone Therapy Followed by Copaxone for Multiple Sclerosis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Siyu Liu, VP, NA Innovative R&D, Teva Neuroscience
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NC-100
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Glatiramer Acetate; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Copaxone 20 mg (Active Comparator): Copaxone 20 mg
  Interventions: Drug: glatiramer acetate 20 mg
- Copaxone 20mg with Novantrone induction (Active Comparator): Copaxone 20mg with Novantrone induction
  Interventions: Drug: glatiramer acetate 20 mg, with mitoxantrone

INTERVENTIONS:
Drug: glatiramer acetate 20 mg — glatiramer acetate 20 mg
  Other Names: Copaxone
  Arms: Copaxone 20 mg
Drug: glatiramer acetate 20 mg, with mitoxantrone — glatiramer acetate 20 mg, with mitoxantrone
  Other Names: Copaxone, Novantrone
  Arms: Copaxone 20mg with Novantrone induction

SUMMARY:
It is thought that treating multiple sclerosis with Novantrone for a short period of time prior to treatment with Copaxone may enhance the onset effect of Copaxone.

ELIGIBILITY:
Inclusion Criteria:

1. Definite MS as determined by the McDonald criteria (Ann Neurol, July 2001) with a relapsing disease course.
2. 2.EDSS 0.0 - 6.5 inclusive
3. 18 to 55 years of age
4. 1 or more T1 Gadolinium-enhancing lesions but no more than 15 lesions
5. Able and willing to sign and date an informed consent form

Exclusion Criteria:

1. Patients ever treated with Glatiramer Acetate or Mitoxantrone.
2. Patients treated with interferons or IV immunoglobulins (IV Ig) in the previous 4 weeks prior to screening visits.
3. Patients treated with methotrexate or azathioprine in the previous 6 months prior to screening visits.
4. Patients ever treated with cyclophosphamide or Total Lymphoid Irradiation (TLI), or cladribine for injection or anthracenediones or anthracyclines, or prior mediastinal radiotherapy.
5. Patients treated with intravenous or oral steroids within 28 days prior to initial MRI.
6. Female patients must be non-pregnant, non-lactating, have a negative screening pregnancy test, and must use contraceptive methods deemed reliable by the investigator.
7. Male patients and their partners must use contraceptive methods deemed reliable by the investigator
8. LVEF < 50%
9. Patients using catheters or Foley catheters
10. Patients who have any other known significant systemic medical disease which may confound the evaluation of the study results such as: ALS, cervical spondylitic myelopathy, syphilis, arteritis, cerebellar syndrome (i.e., due to heredodegeneration), B12/folate deficiency, lyme disease, HTLV 1-myelopathy
11. Patients with immune deficiency or other medical condition that would preclude treatment with Mitoxantrone or Glatiramer Acetate
12. Abnormal screening blood tests exceeding any of the limits defined below:

    Alanine transaminase (ALT) - twice the upper limit of normal Aspartate transaminase (AST) - twice the upper limit of normal Total white blood cell count < 2.3 x 103/uL Baseline neutrophil counts of < 1.5 x103/uL Platelet count < 80 x 103/uL Creatinine >1.5 mg/dL Prothrombin time greater than 150% upper limit of normal
13. Patients with any medical or psychiatric conditions that would make the patient unsuitable for this research, as determined by the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2003-06; Primary Completion 2005-01 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Determine if short-term immunosuppression with mitoxantrone (Novantrone®) followed by chronic treatment with Glatiramer Acetate (GA) in comparison to treatment with GA for the same period of time but without immunosuppression is well-tolerated and safe | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Siyu Liu, MD, Study Director — Teva Neuroscience, Inc.